CLINICAL TRIAL: NCT01925833
Title: Comparison of Adenoma Detection by Polypectomy During Both Insertion and Withdrawal Versus Only Withdrawal of Colonoscopy: a Randomized, Controlled Trial
Brief Title: Adenoma Detection by Polypectomy During Both Insertion and Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong-Seon Ji, Dr, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Insertion
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Adenoma of Large Intestine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Both insertion and withdrawal (Experimental)
  Interventions: Procedure: Both insertion and withdrawal
- Only withdrawal (Active Comparator)
  Interventions: Procedure: Only withdrawal

INTERVENTIONS:
Procedure: Both insertion and withdrawal — inspection and polypectomy during both insertion and withdrawal of colonoscopy
  Arms: Both insertion and withdrawal
Procedure: Only withdrawal — inspection and polypectomy during only withdrawal of colonoscopy
  Arms: Only withdrawal

SUMMARY:
Standard method of colonoscopy is to insert the colonoscope rapidly to reach the cecum, with careful inspection and polypectomy during the withdrawal phase. However, small polyps (e.g. <1cm) seen during insertion phase are difficult to find during withdrawal phase. Also, colon is in different conformation during insertion and withdrawal phases. We think careful inspection and polypectomy during both insertion and withdrawal can improve adenoma detection rate.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing screening or surveillance colonoscopy

Exclusion Criteria:

* Previous colorectal resection, Polyposis syndrome, Inflammatory bowel disease

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1142 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 4 weeks

SECONDARY OUTCOMES:
Number of adenoma per patient | 4 weeks

OTHER OUTCOMES:
Polyp miss rate | 4 weeks

REFERENCES:
- [Derived] Gweon TG, Lee SW, Ji JS, Lee JR, Kim JS, Kim BW, Choi H. Comparison of adenoma detection by colonoscopy between polypectomy performed during both insertion and withdrawal versus during withdrawal only: a multicenter, randomized, controlled trial. Surg Endosc. 2020 Dec;34(12):5461-5468. doi: 10.1007/s00464-019-07342-4. Epub 2020 Jan 17. PMID 31953727